CLINICAL TRIAL: NCT06398613
Title: Preoperative PSMA PET/CT As Triage for Extended Pelvic Lymph Node Dissection (ePLND) in Patients Scheduled for Robot-Assisted Laparoscopic Radical Prostatectomy (RALP)
Brief Title: Preoperative PSMA PET/CT As Triage for EPLND in Patients Scheduled for RALP (PrePSMA)
Acronym: PrePSMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Viktor Berge, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK 688379
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: PSMA PET/CT, ePLND
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RALP + ePLND Arm A (No Intervention): RALP + ePLND
- RALP +/- ePLND Arm B (Experimental): I preoperative PSMA PET/CT is positive for pelvic nodal metastasis, ePLND concomitant with RALP will be performed. If PSMA PET/CT is negative, only RALP will be done.
  Interventions: Diagnostic Test: extended pelvic lymph node dissection (ePLND)

INTERVENTIONS:
Diagnostic Test: extended pelvic lymph node dissection (ePLND) — Prostate-Specific Membrane Antigen Emission Tomography/Computed Tomography (PSMA PET/CT) will done preoperatively in both arms of the study. In arm A all patients will undergo ePLND, in arm B only patients with positive PSMA PET/CT will undergo ePLND
  Arms: RALP +/- ePLND Arm B

SUMMARY:
Extended pelvic lymph node dissection (ePLND) is considered the gold standard for nodal staging in men with prostate cancer (PCa). The aim of this project is to determine if preoperative prostate specific membrane antigen (PSMA) positron emission tomography (PET)/computed tomograpy (CT) can safely replace ePLND as a staging method in PCa patients undergoing robot-assisted laparoscopic radical prostatectomy (RALP).

DETAILED DESCRIPTION:
Due to the latest change in EAU guidelines in May 2024, all eligible patients will undergo PSMA PET/CT. Patients will then be randomized between RALP and ePLND (Arm A) and RALP +/- ePLND (arm B): If PSMA PET/CT detect suspicious pelvic nodes, the patient will undergo ePLND concomitant with RALP. If PSMA PET/CT is negative, only RALP will be performed .

Primary outcome measures:

Difference in biochemical recurrence (BCR) rate between arm A and arm B within 2 years after initiation of primary treatment (BCR ≥ 0.2 ng/ml).

Secondary outcome measures:

Difference between Arm A and Arm B for surgical complications, persistent PSA after RALP and initiation of salvage therapy

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven diagnosed adenocarcinoma of the prostate
* Indication for ePLND combined with RALP:
* High-risk group (EAU) and including MRI findings indicating extra prostatic extension (Likert scale ≥4)
* -ISUP GG 3 with ≥1 of the following unfavourable risk factors

  * cT2b-c,
  * ≥50% percentage of positive biopsy cores,
  * PSA 10-20
* cN1 selected to surgery
* Written informed consent
* No known allergies for PSMA tracer
* 18 years and older

Exclusion Criteria:

* History of previously actively treated PCa
* Previous malignancies (except basal cell carcinoma of the skin) that has not been recurrence-free past ≥5 years
* Unwillingness or inability to undergo PSMA PET/CT and/or ePLND and RALP
* Presence of distant metastasis (cM1) on MRI imaging

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between Arm A and Arm B in biochemical recurrence (BCR) rate between groups within 2 years after initiation of RALP | 2 years after initiation of primary treatment
  BCR is defined as PSA ≥ 0.2 ng/ml

SECONDARY OUTCOMES:
Difference between Arm A and Arm B in incidence and types of surgical complications | 3 months follow up
  Clavien Dindo classification of complications will be used
Difference between Arm A and Arm B in persistent PSA after RALP | 2 months after RALP
  If the PSA value 6 weeks postoperatively is > 0.10 ng/ml the patient has persistent PSA
Difference between Arm A and Arm B in initiation of salvage therapy | 2 years follow up
  Salvage therapy is salvage radiation therapy, salvage surgery and ADT

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Berge, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway